CLINICAL TRIAL: NCT05517330
Title: Neoadjuvant Tislelizumab With Afatinib for the Treatment of Resectable Head and Neck Squamous Cell Carcinoma: A Single-Arm Phase 2 Trial (neoCHANCE-1 Trial)
Brief Title: Neoadjuvant Tislelizumab With Afatinib for Resectable Head and Neck Squamous Cell Carcinoma
Acronym: neoCHANCE-1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Xingchen Peng, Professor, West China Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ChiECRCT20210619
Record Dates: First submitted 2022-08-19; First posted 2022-08-26 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Head and Neck Cancer
Keywords: Head and Neck Cancer; Neoadjuvant therapy; Immunotherapy; EGFR-TKI
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — tislelizumab; Afatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment Cohort (Experimental): * Tislelizumab administration on days 1 and 22, and afatinib continuous administration from days 1 to 42
  * Standard of care surgery
  Interventions: Biological: Tislelizumab; Drug: Afatinib

INTERVENTIONS:
Biological: Tislelizumab — 200mg IV Q3W
  Other Names: BGB-A317
Drug: Afatinib — 30mg PO QD

SUMMARY:
The purpose of this study is to explore the efficiency and safety of anti-Programmed death-1 (PD-1) immunotherapy, tislelizumab, combined with EGFR-tyrosine kinase inhibitor (TKI), afatinib as a new neoadjuvant treatment regimen for patients with resectable head and neck squamous cell carcinoma (HNSCC).

DETAILED DESCRIPTION:
Head and neck squamous cell carcinoma (HNSCC) is the most common malignancy of the head and neck. More than 60% of patients with HNSCC have locally advanced or metastatic disease at the time of diagnosis, with a 5-year overall survival rate of less than 60%. The clinical outcomes of those patients still need to be improved.

Neoadjuvant therapy theoretically can reduce tumor volume, increase organ retention rate, and reduce distant metastasis rate. However, in addition to nasopharyngeal carcinoma, results from several phase III clinical trials have not proved a significant survival benefit of neoadjuvant chemotherapy for patients with resectable HNSCC. It is urgent to explore new neoadjuvant treatment options to improve the prognosis of patients with HNSCC.

Immunotherapy such as PD-1/PD-L1 inhibitors have shown excellent efficiency in the treatment of malignancies. Anti-PD-1 therapy is approved as the first-line treatment of recurrent/metastatic HNSCC. Neoadjuvant immunotherapy for the treatment of locally advanced and resectable HNSCC has been demonstrated to be feasible in some trials.

Afatinib, as an irreversible ErbB tyrosine kinase inhibitor (TKI), has been used as the second-line treatment for recurrent and/or metastatic HNSCC. However, there is a lack of high-level evidence-based medical evidence for the use of afatinib in preoperative therapy for HNSCC. A previous study published in 2018 confirmed that afatinib can be administered safely before surgery.

In summary, the investigators designed this study to explore the efficiency and safety of anti-PD1 immunotherapy, tislelizumab, combined with EGFR-TKI, afatinib as a new neoadjuvant treatment regimen for patients with resectable HNSCC, aiming to provide a new treatment option for those patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or above.
2. Patients with pathologically confirmed HNSCC (except for nasopharyngeal carcinoma) and meet the following conditions:

   * were newly diagnosed and without distant metastasis;
   * were deemed surgically resectable evaluated by a head and neck surgeon;
   * were willing to undergo surgery.
3. Eastern Cooperative Oncology Group (ECOG) performance status 0-1.
4. Adequate organ and bone marrow function:

   * absolute neutrophil count ≥ 1.5 × 10^9/L, hemoglobin ≥ 80 g/L, platelets ≥ 80 × 10^9/L;
   * ALT, AST and ALP < 2.5× upper limit of normal (ULN), total bilirubin ≤ 2×ULN; albumin≥ 2.8 g/dL；
   * creatinine clearance ≥ 60 ml/min；
   * INR≤ 1.5, APTT≤ 1.5×ULN.
5. Written informed consent.

Exclusion Criteria:

1. History of other malignancies (except for the history of malignant tumors that have been cured and have not recurred within 5 years, such as skin basal cell carcinoma, skin squamous cell carcinoma, superficial bladder cancer, in situ cervical cancer, and gastrointestinal mucosal cancer, etc.）
2. Have an active autoimmune disease requiring systemic treatment or a documented history of clinically severe autoimmune disease.
3. Any history of allergic disease, or a sever hypersensitivity reaction to drugs, or allergy to the study drug components.
4. Any of prior therapy with:

   * anti-PD-1, anti-PD-L1/2, anti-CTLA-4 antibody, anti-EGFR antibody or EGFR-TKIs；
   * antitumor vaccine;
   * any active vaccine against an infectious disease within 4 weeks prior to the first dose or planned during the study period;
   * major surgery or serious trauma within 4 weeks before the first dose;
   * toxicity from prior antitumor therapy has not recovered to ≤ CTCAE Version 5.0 Grade 1 or the level specified by the inclusion/exclusion criteria.
5. With serious medical diseases, such as grade II and above cardiac dysfunction (NYHA criteria), ischemic heart disease, supraventricular or ventricular arrhythmia, poorly controlled diabetes mellitus, poorly controlled hypertension, echocardiographic ejection fraction < 50%, etc.
6. With interstitial pneumonitis, non-infectious pneumonitis, active pulmonary tuberculosis, or history of pulmonary tuberculosis infection that were not controlled by treatment.
7. With hyperthyroidism, or organic thyroid disease.
8. With active infection, or unexplained fever during the screening period or 48 hours before the first dose.
9. With active hepatitis B or C, or known history of positive HIV test, or acquired immunodeficiency syndrome.
10. History of a clear neurological or psychiatric disorder.
11. History of drug abuse or alcohol abuse.
12. Women who are pregnant or breastfeeding, or have a reproductive plan from the screening period to 3 months after the end of the study, or have sex without contraceptive measures, or are unwilling to take appropriate contraceptive measures.
13. Received any investigational drug within 4 weeks prior to the first dose, or concurrently enrolled in another clinical trial.
14. Any other factors that are not suitable for inclusion in this study judged by investigators.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2022-09-19 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
Major Pathologic Response | Time of surgery
  Major Pathologic Response (MPR) was defined as fewer than 10% viable tumor cells.

SECONDARY OUTCOMES:
Pathologic Complete Response | Time of surgery
  Pathologic Complete Response (pCR) was defined as the absence of viable tumor cells.
Objective Response Rate | Up to 8 weeks
  Objective Response Rate (ORR) was defined as the percentage of participants with a best overall response of CR or PR using RECIST Criteria.
Adverse events | Up to 12 weeks
  Adverse events were defined as the number of participants with adverse events using CTCAE Criteria or with an unplanned surgery delay.
Disease-free Survival | 1 year
  Disease-free Survival (DFS) was defined as the time from the administration of the first dose to first disease progression or death.

CONTACTS AND LOCATIONS:
Overall Officials: Xingchen Peng, Professor, Principal Investigator — West China Hospital
Locations (1):
- Xingchen Peng, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ferlay J, Colombet M, Soerjomataram I, Mathers C, Parkin DM, Pineros M, Znaor A, Bray F. Estimating the global cancer incidence and mortality in 2018: GLOBOCAN sources and methods. Int J Cancer. 2019 Apr 15;144(8):1941-1953. doi: 10.1002/ijc.31937. Epub 2018 Dec 6. PMID 30350310
- [Background] Bray F, Ferlay J, Soerjomataram I, Siegel RL, Torre LA, Jemal A. Global cancer statistics 2018: GLOBOCAN estimates of incidence and mortality worldwide for 36 cancers in 185 countries. CA Cancer J Clin. 2018 Nov;68(6):394-424. doi: 10.3322/caac.21492. Epub 2018 Sep 12. PMID 30207593
- [Background] Pulte D, Brenner H. Changes in survival in head and neck cancers in the late 20th and early 21st century: a period analysis. Oncologist. 2010;15(9):994-1001. doi: 10.1634/theoncologist.2009-0289. Epub 2010 Aug 26. PMID 20798198
- [Background] Denaro N, Merlano MC, Russi EG. Follow-up in Head and Neck Cancer: Do More Does It Mean Do Better? A Systematic Review and Our Proposal Based on Our Experience. Clin Exp Otorhinolaryngol. 2016 Dec;9(4):287-297. doi: 10.21053/ceo.2015.00976. Epub 2016 Jun 25. PMID 27337948
- [Background] Harari PM. Promising new advances in head and neck radiotherapy. Ann Oncol. 2005;16 Suppl 6:vi13-vi19. doi: 10.1093/annonc/mdi453. PMID 15987991
- [Background] Haddad R, O'Neill A, Rabinowits G, Tishler R, Khuri F, Adkins D, Clark J, Sarlis N, Lorch J, Beitler JJ, Limaye S, Riley S, Posner M. Induction chemotherapy followed by concurrent chemoradiotherapy (sequential chemoradiotherapy) versus concurrent chemoradiotherapy alone in locally advanced head and neck cancer (PARADIGM): a randomised phase 3 trial. Lancet Oncol. 2013 Mar;14(3):257-64. doi: 10.1016/S1470-2045(13)70011-1. Epub 2013 Feb 13. PMID 23414589
- [Background] Cohen EE, Karrison TG, Kocherginsky M, Mueller J, Egan R, Huang CH, Brockstein BE, Agulnik MB, Mittal BB, Yunus F, Samant S, Raez LE, Mehra R, Kumar P, Ondrey F, Marchand P, Braegas B, Seiwert TY, Villaflor VM, Haraf DJ, Vokes EE. Phase III randomized trial of induction chemotherapy in patients with N2 or N3 locally advanced head and neck cancer. J Clin Oncol. 2014 Sep 1;32(25):2735-43. doi: 10.1200/JCO.2013.54.6309. Epub 2014 Jul 21. PMID 25049329
- [Background] Geoffrois L, Martin L, De Raucourt D, Sun XS, Tao Y, Maingon P, Buffet J, Pointreau Y, Sire C, Tuchais C, Babin E, Coutte A, Rolland F, Kaminsky MC, Alfonsi M, Lapeyre M, Saliou M, Lafond C, Jadaud E, Gery B, Zawadi A, Tourani JM, Khoury C, Henry AR, Hasbini A, Guichard F, Borel C, Meert N, Guillet P, Calais MH, Garaud P, Bourhis J. Induction Chemotherapy Followed by Cetuximab Radiotherapy Is Not Superior to Concurrent Chemoradiotherapy for Head and Neck Carcinomas: Results of the GORTEC 2007-02 Phase III Randomized Trial. J Clin Oncol. 2018 Nov 1;36(31):3077-3083. doi: 10.1200/JCO.2017.76.2591. Epub 2018 Jul 17. PMID 30016178
- [Background] Ferris RL, Blumenschein G Jr, Fayette J, Guigay J, Colevas AD, Licitra L, Harrington K, Kasper S, Vokes EE, Even C, Worden F, Saba NF, Iglesias Docampo LC, Haddad R, Rordorf T, Kiyota N, Tahara M, Monga M, Lynch M, Geese WJ, Kopit J, Shaw JW, Gillison ML. Nivolumab for Recurrent Squamous-Cell Carcinoma of the Head and Neck. N Engl J Med. 2016 Nov 10;375(19):1856-1867. doi: 10.1056/NEJMoa1602252. Epub 2016 Oct 8. PMID 27718784
- [Background] Burtness B, Harrington KJ, Greil R, Soulieres D, Tahara M, de Castro G Jr, Psyrri A, Baste N, Neupane P, Bratland A, Fuereder T, Hughes BGM, Mesia R, Ngamphaiboon N, Rordorf T, Wan Ishak WZ, Hong RL, Gonzalez Mendoza R, Roy A, Zhang Y, Gumuscu B, Cheng JD, Jin F, Rischin D; KEYNOTE-048 Investigators. Pembrolizumab alone or with chemotherapy versus cetuximab with chemotherapy for recurrent or metastatic squamous cell carcinoma of the head and neck (KEYNOTE-048): a randomised, open-label, phase 3 study. Lancet. 2019 Nov 23;394(10212):1915-1928. doi: 10.1016/S0140-6736(19)32591-7. Epub 2019 Nov 1. PMID 31679945
- [Background] Machiels JP, Haddad RI, Fayette J, Licitra LF, Tahara M, Vermorken JB, Clement PM, Gauler T, Cupissol D, Grau JJ, Guigay J, Caponigro F, de Castro G Jr, de Souza Viana L, Keilholz U, Del Campo JM, Cong XJ, Ehrnrooth E, Cohen EE; LUX-H&N 1 investigators. Afatinib versus methotrexate as second-line treatment in patients with recurrent or metastatic squamous-cell carcinoma of the head and neck progressing on or after platinum-based therapy (LUX-Head & Neck 1): an open-label, randomised phase 3 trial. Lancet Oncol. 2015 May;16(5):583-94. doi: 10.1016/S1470-2045(15)70124-5. Epub 2015 Apr 16. PMID 25892145
- [Background] Guo Y, Ahn MJ, Chan A, Wang CH, Kang JH, Kim SB, Bello M, Arora RS, Zhang Q, He X, Li P, Dechaphunkul A, Kumar V, Kamble K, Li W, Kandil A, Cohen EEW, Geng Y, Zografos E, Tang PZ. Afatinib versus methotrexate as second-line treatment in Asian patients with recurrent or metastatic squamous cell carcinoma of the head and neck progressing on or after platinum-based therapy (LUX-Head & Neck 3): an open-label, randomised phase III trial. Ann Oncol. 2019 Nov 1;30(11):1831-1839. doi: 10.1093/annonc/mdz388. PMID 31501887
- [Background] Burtness B, Haddad R, Dinis J, Trigo J, Yokota T, de Souza Viana L, Romanov I, Vermorken J, Bourhis J, Tahara M, Martins Segalla JG, Psyrri A, Vasilevskaya I, Nangia CS, Chaves-Conde M, Kiyota N, Homma A, Holeckova P, Del Campo JM, Asarawala N, Nicolau UR, Rauch D, Even C, Wang B, Gibson N, Ehrnrooth E, Harrington K, Cohen EEW; LUX-Head & Neck 2 investigators. Afatinib vs Placebo as Adjuvant Therapy After Chemoradiotherapy in Squamous Cell Carcinoma of the Head and Neck: A Randomized Clinical Trial. JAMA Oncol. 2019 Aug 1;5(8):1170-1180. doi: 10.1001/jamaoncol.2019.1146. PMID 31194247
- [Background] Machiels JP, Bossi P, Menis J, Lia M, Fortpied C, Liu Y, Lhommel R, Lemort M, Schmitz S, Canevari S, De Cecco L, Guzzo M, Bianchi R, Quattrone P, Crippa F, Duprez T, Lalami Y, Quiriny M, de Saint Aubain N, Clement PM, Coropciuc R, Hauben E, Licitra LF. Activity and safety of afatinib in a window preoperative EORTC study in patients with squamous cell carcinoma of the head and neck (SCCHN). Ann Oncol. 2018 Apr 1;29(4):985-991. doi: 10.1093/annonc/mdy013. PMID 29346507